CLINICAL TRIAL: NCT02562833
Title: The PLE²NO Self-management and Exercise Program for Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: The PLE²NO Self-management and Exercise Program for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Lisbon (Other)
Responsible Party: Principal Investigator, Priscila Marconcin, Master degree, Technical University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PLENO-FMH-1
Record Dates: First submitted 2015-09-23; First posted 2015-09-29 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Self-management; Multi-Component Exercise
MeSH Terms: conditions — Osteoarthritis | interventions — Exercise Therapy; Models, Educational

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-Management and exercise (Experimental)
  Interventions: Device: Self-Management and exercise
- Educational (Active Comparator)
  Interventions: Device: Educational

INTERVENTIONS:
Device: Self-Management and exercise — Self-Management and exercise It is a 3 months intervention where the participants were enrolled two times per week, 90 minutes each session, first 30 minutes were allocated for the self-management component and the remaining 60 minutes for the exercise component. Additionally,participants received glucosamine and chondroitin sulfate supplement.
  Arms: Self-Management and exercise
Device: Educational — This group received an educational book with information about OA features, treatment modalities and exercise education with illustration. Additionally, a monthly educational session each with one hour and a half duration, in total 3, where joint protections strategies, OA self-management and exercise contents were transmitted. Additionally,participants received glucosamine and chondroitin sulfate supplement.
  Arms: Educational

SUMMARY:
The PLE²NO (in Portuguese Education and Exercise Free Program for osteoarthritis) is a self-management and exercise program specific for elderly with knee osteoarthritis (OA), with the goals of managing OA symptoms, improving physical fitness, and developing self-efficacy and self-management of pathology.

DETAILED DESCRIPTION:
Participants were randomly assigned to one of two groups: (1) Self-management and Exercise (2) Educational. Both groups received glucosamine and chondroitin sulfate supplement during the intervention. Blinding of participants was not possible due to the nature of the intervention; however, assessors were blinded to group allocation. The PLE2NO (in Portuguese Education and Exercise Free Program for osteoarthritis) is a community-based program with two components: self-management and exercise. Each session lasted 90 minutes, and the first 30 minutes corresponded to a self-management part and the remaining 60 minutes to the exercise program. The program was offered in a group format, encouraging peer interactions and socialization that can help counteract feelings of depression and isolation. The self-management program is based on the program developed at Stanford University, the Chronic Disease Self-Management Program which the purpose is developing self-efficacy based on social cognitive theory. The exercise program comprised both health related (strength, flexibility) and skill-related (agility, balance, speed and power) physical fitness components, and was based on Fit an Strong Program, on Exercise for People with Arthritis (FEPA) and also on the program Takin Control with Exercise (Arthritis Foundation). The program will last for 3 months and 6 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age over than or equal to 60 years;
2. Bilateral or unilateral OA of the knee diagnosed according to clinical and radiological criteria of the American College of Rheumatology (ACR)(Altman et al., 1986);
3. Independent mobility;
4. and reading and writing knowledge.

Exclusion Criteria:

1. Not be involved in another intervention program (exercise, education or physical therapy;
2. Do not use supplements (chondroitin sulfate and / or glucosamine) for at least three months;
3. Have other pathology (cardiovascular, respiratory, musculoskeletal, cancer) that prevents physical exercise;
4. Mental / psychological state hindering understanding of the program;
5. Having undergone surgery for knee replacement or going perform this surgery in the next eight months;
6. Being allergic to shellfish;
7. Have made injections of corticosteroids or hyaluronic acid in the last 6 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-02; Primary Completion 2015-02 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline knee OA symptoms to 3 month, assessed by Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire. | Change from baseline to 3 month
Change from baseline self-efficacy to 3 month, assessed by Self-efficacy for managing Chronic Disease - 6-Item Scale questionnaire. | Change from baseline to 3 month
Change from baseline functional strength to 3 month, assessed by Five repetition sit to stand test. | Change from baseline to 3 month
Change from baseline cardiorespiratory endurance to 3 month, assessed by Six Minutes' Walk test. | Change from baseline to 3 month
Change from baseline flexibility to 3 month, assessed by Chair Sit and Reach test, and the Back Scratch test. | Change from baseline to 3 month
Change from baseline hand grip strength to 3 month, assessed by hand grip dynamometer test. | Change from baseline to 3 month

SECONDARY OUTCOMES:
Change from baseline health related quality of life to 3 month, assessed by perception of health and quality of life five dimension, five levels (EuroQol - EQ-5D-5L) questionnaire. | Change from baseline to 3 month
Change from baseline self-management behaviors to 3 month, Use of cognitive symptom management techniques, Communication with Physicians questionnaires. | Change from baseline to 3 month
Change from baseline physical activity level to 3 month, assessed by International Physical Activity Questionnaire (IPAQ). | Change from baseline to 3 month
Change from baseline gait speed to 3 month, assessed by Six-meters test. | Change from baseline to 3 month
Change from baseline balance to 3 month, assessed by Standing Balance test. | Change from baseline to 3 month
Change from baseline mobility to 3 month, assessed by Timed "up-and-go" test. | Change from baseline to 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Priscila Marconcin, Master, Principal Investigator — Faculty of Human Kinetics, Lisbon University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Marconcin P, Espanha M, Yazigi F, Campos P. The PLE(2)NO self-management and exercise program for knee osteoarthritis: Study Protocol for a Randomized Controlled Trial. BMC Musculoskelet Disord. 2016 Jun 7;17:250. doi: 10.1186/s12891-016-1115-7. PMID 27267755